CLINICAL TRIAL: NCT03615157
Title: Effects of a Home-based Exercise Program on Functional Capacity and Quality of Life in Heart Failure Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other); InCor Heart Institute (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, NAOMI KONDO NAKAGAWA NAOMI KONDO, Associate Professor of Medical School of Sao Paulo University, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 411/14
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Chronic Heart Failure
Keywords: Home-based exercise; Functional capacity; Chronic Heart Failure
MeSH Terms: interventions — Exercise Therapy; Resistance Training

STUDY DESIGN:
Intervention Model Description: The participants will be randomized in two groups: Home-based and Supervised exercise groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based exercise rehabilitation (Experimental): Patients will be submitted to a 12-weeks training program, with walking at 60-70% of heart rate reserve monitored by a heart rate monitor (30 minutes/session for 5 days/week) and peripheral muscle training including upper and lower limbs (50% of the 1-maximum repetition test)
  Interventions: Other: Exercise rehabilitation
- Supervised exercise rehabilitation (Active Comparator): Patients will be submitted to a 12-weeks training program, with sessions (3 days/week) supervised by a physiotherapist, including cycling at 60-70% of heart rate reserve and peripheral muscle training of upper and lower limbs (50% of the 1-maximum repetition test)
  Interventions: Other: Exercise rehabilitation

INTERVENTIONS:
Other: Exercise rehabilitation — Patients will be submitted to a twelve-week combined exercise program of aerobic and peripheral muscle training. They will be randomized in two groups: Home-based and Supervised.
  Other Names: Aerobic and resistance training

SUMMARY:
Heart failure (HF) is a multisystemic disease leading to exercise intolerance and fatigue. Supervised physical training improves functional capacity, quality of life and reduces hospital admissions in HF patients. In this way, home physical training may be a good alternative to patients who, for any reason, cannot perform supervised training. Objective: To asses the effects of a home-based training program on functional capacity, sedentary lifestyle and quality of life of patients with chronic HF compared to supervised training.

DETAILED DESCRIPTION:
After agreement with the written informed consent, subjects with heart failure (left ventricle ejection fraction bellow or equal 40%) will be included in this study. They will be randomized in two groups: Home-based and Supervised exercise groups. The two groups will be submitted to a twelve-week combined exercise program of aerobic and peripheral muscle training. All volunteers will be assessed at baseline and after twelve weeks of intervention. Peripheric and respiratory muscle strength as well the 6MW analyses were assessed also at 4 and 8 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure (functional class from NYHA II and III),
* Left ventricle ejection fraction bellow or equal to 40%
* Clinical stability during the last three months
* Medical release for physical training after cardiopulmonary test

Exclusion Criteria:

* Uncontrolled arrhythmia
* Pulmonary artery systolic pressure > 35 mmHg by the echo doppler cardiogram,
* Peripheral oxygen saturation < 92% in resting condition
* Respiratory infection in the previous 30 days to the enrollment into the study
* Cognitive, neurological or orthopedic limitations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-02-15 (Estimated)

PRIMARY OUTCOMES:
Changes in peak oxygen uptake (ml/kg/min) | Baseline and after 12 weeks of exercise programs
  Patients will be submitted to cardiopulmonary treadmill exercise tests at baseline and after 12 weeks.

SECONDARY OUTCOMES:
Incidence of cardiac events and arrhythmia | Baseline and after 12 weeks of exercise programs
  By a 24-hours holter system for continuous recording of ambulatory electrocardiographic signs
Changes in distance from the six minute walk test (6MW, m) | Baseline and after 4, 8 and 12 weeks of exercise programs
  Patients will be submitted to the 6MW accordingly to the American Thoracic guidelines to assess functional capacity using the six minute walk test
Changes in respiratory muscle strength (cmH2O) | Baseline and after 4, 8 and 12 weeks of exercise programs
  Inspiratory and expiratory muscle strength will be assessed using an analogic pressure transducer
Changes in peripheral muscle strength (N) - Quadriceps mm | Baseline and after 4, 8 and 12 weeks of exercise program
  Quadriceps strength will be assessed by MicroFet 2 dynamometer (HogganHealth, USA)
Changes in peripheral muscle strength (kgf) - Hand grip | Baseline and after 4, 8 and 12 weeks of exercise programs
  Hand grip strength will be assessed by Jamar dynamometer (Sammons Preston Rolyan, 4, Sammons Court, Bolingbrook, IL, 60440)
Changes in daily physical activity and sedentary lifestyle | Baseline and after 12 weeks of exercise programs
  Patients will use the accelerometer GT3X (Actigraph, Pensacola, FL, USA) on waist during 9 days to asses daily physical activity and sedentary lifestyle
Changes in International Physical Activity Questionnaire (IPAQ) | Baseline and after 12 weeks of exercise programs
  Patients will be classified as sedentary, irregularly active, active or very active according to Matsudo's Classification (2001)
Changes in quality of life using SF-36 | Baseline and after 12 weeks of exercise programs
  Quality of life will be assessed by the Short Form-36 Questionnaire
Changes in quality of life using MLHF | Baseline and after 12 weeks of exercise programs
  Quality of life will be assessed by the Minnesota Living with Heart Failure Questionnaire
Changes in brain natriuretic peptide (BNP, pg/mL) | Baseline and after 12 weeks of exercise programs
  A blood sample of 5 ml will be collected in a tube and BNP will be measured
Changes in heart rate variability (HRV) | Baseline and after 12 weeks of exercise programs
  HRV will be analysed from the spectral analysis of R-R intervals obtained from a heart rate monitor (Polar, S810, Kempele, Finland) during the 6MW
Changes in sleep quality | Baseline and after 12 weeks of exercise programs
  Patients will use the accelerometer GT3X (Actigraph, Pensacola, FL, USA) on wrist for nine days to asses Sleep quality. Furthermore, the Pittsburgh Sleep Quality Index will be used to classify patients as good or poor sleepers.
Changes in daytime sleepiness | Baseline and after 12 weeks of exercise programs
  Daytime sleepiness will be assessed by the Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - School of Medicine, University of Sao Paulo, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
we will insert all individual data in a common website for research
Supporting Information: Study Protocol, CSR
Time Frame: As soon as we have half data, we will make that available
Access Criteria: For researchers

REFERENCES:
- [Derived] Andrade GN, Umeda IIK, Fuchs ARCN, Mastrocola LE, Rossi-Neto JM, Moreira DAR, Oliveira PA, Andre CDS, Cahalin LP, Nakagawa NK. Home-based training program in patients with chronic heart failure and reduced ejection fraction: a randomized pilot study. Clinics (Sao Paulo). 2021 Jun 11;76:e2550. doi: 10.6061/clinics/2021/e2550. eCollection 2021. PMID 34133657